CLINICAL TRIAL: NCT01049360
Title: Efficacy and Safety Study of Two Fixed-Dose Combinations of Aclidinium Bromide With Formoterol Fumarate Compared With Aclidinium Bromide, Formoterol Fumarate, and Placebo All Administered Twice Daily (BID) to Patients With Stable, Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Study of Two Fixed-dose Combinations of Aclidinium Bromide With Formoterol Fumarate Compared With Aclidinium Bromide, Formoterol Fumarate and Placebo
Acronym: LAC-MD-27
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAC-MD-27
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Aclidinium 400 μg / Formoterol 12 μg (Experimental): Aclidinium bromide 400 μg / formoterol fumarate 12 μg fixed dose combination administered twice-daily (BID)
  Interventions: Drug: Aclidinium 400 μg / Formoterol 12 μg
- Aclidinium 400 μg / formoterol 6 μg (Experimental): Aclidinium bromide 400 μg / formoterol fumarate 6 μg fixed dose combination administered twice-daily (BID)
  Interventions: Drug: Aclidinium 400 μg / Formoterol 6 μg
- Aclidinium 400 μg (Experimental): Aclidinium bromide 400 μg administered twice-daily (BID)
  Interventions: Drug: Aclidinium 400 μg
- Formoterol 12 μg (Active Comparator): Formoterol fumarate 12 μg twice-daily
  Interventions: Drug: Formoterol 12 μg
- Placebo (Placebo Comparator): Placebo twice-daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium 400 μg / Formoterol 12 μg — Aclidinium bromide 400 μg / formoterol fumarate 12 μg fixed dose combination administered twice-daily (BID) for a 14 day period within four different treatment periods.
  Arms: Aclidinium 400 μg / Formoterol 12 μg
Drug: Aclidinium 400 μg / Formoterol 6 μg — Aclidinium bromide 400 μg / formoterol fumarate 6 μg fixed dose combination administered twice-daily (BID) for a 14 day period within four different treatment periods.
  Arms: Aclidinium 400 μg / formoterol 6 μg
Drug: Aclidinium 400 μg — Aclidinium bromide 400 μg administered twice-daily (BID) for a 14 day period within four different treatment periods.
  Arms: Aclidinium 400 μg
Drug: Formoterol 12 μg — Formoterol fumarate 12 μg twice-daily for a 14 day period within four different treatment periods.
  Arms: Formoterol 12 μg
Drug: Placebo — Placebo twice-daily delivered by inhalation for a 14 day period within four different treatment periods.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of this multicenter, randomized, double-blind, placebo-controlled, 4-period, incomplete-block crossover, dose-ranging study comparing 2 fixed dose combinations (FDCs) of aclidinium bromide with formoterol fumarate or with placebo, aclidinium bromide and formoterol fumarate, all administered twice a day (BID) in patients with stable, moderate to severe chronic obstructive pulmonary disease (COPD) beginning with a 2-week run-in period and with a 7-10 day washout each between treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and be willing to participate in the study as indicated by signing the ICF and HIPAA form
* Be male or female aged 40 to 80 years, inclusive
* Have a diagnosis of stable, moderate to severe COPD (stages II and III) as defined by guidelines of the Global Initiative for Chronic Obstructive Lung Disease (2008)
* Be a current or former cigarette smoker with a smoking history of at least 10 pack-years
* Have post-albuterol/salbutamol FEV1 values ≥ 30% and < 80% of the predicted value. FEV1 will be measured at the Screening Visit (Visit 1) between 10 and 15 minutes after inhalation of albuterol/salbutamol.
* Have post-albuterol/salbutamol FEV1/FVC values < 70% (ie, 100 × post- albuterol/salbutamol FEV1/FVC < 70%).
* If female, be at least 1 year postmenopausal or surgically sterile (defined as having a hysterectomy or tubal ligation). Women of childbearing potential must have a negative serum β-human chorionic gonadotropin pregnancy test at screening
* Be in good stable health (as judged by the Investigator) other than the COPD, based on medical history, physical examination, ECG, spirometry, and clinical laboratory data evaluations
* Have COPD symptoms and FEV1 values at the time of randomization that are stable compared with those at Screening (Visit 1), according to the Investigator's medical judgment

Exclusion Criteria:

* Have been hospitalized for an acute COPD exacerbation within 3 months before screening
* Have any respiratory tract infection (including the upper respiratory tract) or signs of a COPD exacerbation or respiratory infection in the 6 weeks before Screening (Visit 1).
* Have any clinically significant respiratory conditions other than COPD
* Have a history or presence of asthma verified from medical records
* Have used theophylline (including long-acting theophylline) within the previous 3 months before study entry
* Have Stage II hypertension, defined as systolic pressure of 160 and above, and diastolic pressure of 100 and above
* Chronic use of oxygen therapy ≥ 15 hours a day
* Have a history, current diagnosis, or presence of exercise-induced bronchospasm
* Have a body mass index ≥ 40 kg/m2
* Have participated in an pulmonary rehabilitation program within the previous 3 months
* Have clinically significant cardiovascular conditions
* Have uncontrolled infection resulting from human immunodeficiency virus and/or active hepatitis
* Have symptomatic prostatic hypertrophy and/or bladder neck obstruction.
* Have narrow-angle glaucoma
* Have a history of hypersensitivity reaction (including report of paradoxical bronchospasm) to inhaled anticholinergics (including aclidinium bromide), β2 adrenergic agonists, or any other inhaled medication or any component thereof
* Have a QTcB, as indicated in the centralized reading report, above 470 msec in the resting ECGs performed at Screening (Visit 1) and/or patients who are using medications that may prolong the QT interval
* Have clinically relevant abnormalities in the results of clinical laboratory tests, in ECG parameters other than QTc, in results of the physical examination,
* Have any concurrent medical condition that, in the judgment of the Investigator, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
* Do not maintain regular day/night, waking/sleeping cycles (eg, patients with history of sleep apnea syndrome or any disease related with sleep disturbances such as restless legs syndrome or somnambulism)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (20):
- United States (20):
  - Forest Investigative Site 0909, Glendale, Arizona
  - Forest Investigative Site 2050, Pheonix, Arizona
  - Forest Investigative Site 2029, Rancho Mirage, California
  - Forest Investigative Site 1084, Stockton, California
  - Forest Investigative Site 2045, Wheat Ridge, Colorado
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 2053, Tampa, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1431, North Dartmouth, Massachusetts
  - Forest Investigative Site 2084, Summit, New Jersey
  - Forest Investigative Site 1119, Elmira, New York
  - Forest Investigative Site 2035, Elizabeth City, North Carolina
  - Forest Investigative Site 1153, Raleigh, North Carolina
  - Forest Investigative Site 2028, Cincinnati, Ohio
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1106, Portland, Oregon
  - Forest Investigative Site 1089, East Providence, Rhode Island
  - Forest Investigative Site 1121, Spartanburg, South Carolina
  - Forest Investigative Site 1498, San Antonio, Texas
  - Forest Investigative Site 1129, Waco, Texas

REFERENCES:
- See also: lac-md-27-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4066&filename=lac-md-27-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a total of 20 study centers in the United States. The first patient was screened in December 2009 and the last patient visit was in August 2010.
Groups:
- Sequence 1: Aclidiunium/Formoterol 400/6 - Aclidiunium/Formoterol 400/12 - Aclidinium - Formoterol
- Sequence 2: Aclidinium/Formoterol 400/12 - Aclidinium - Formoterol - Placebo
- Sequence 3: Aclidinium - Formoterol - Placebo - Aclidinium/Formoterol 400/6
- Sequence 4: Formoterol - Placebo - Aclidinium/Formoterol 400/6 - Aclidinium/Formoterol 400/12
- Sequence 5: Placebo - Aclidinium/Formoterol 400/6 - Aclidinium/Formoterol 400/12 - Aclidinium
- Sequence 6: Aclidinium/Formoterol 400/6 - Aclidinium - Placebo - Aclidinium/Formoterol 400/12
- Sequence 7: Aclidinium/Formoterol 400/12 - Formoterol - Aclidinium/Formoterol 400/6 - Aclidinium
- Sequence 8: Aclidinium - Placebo - Aclidinium/Formoterol 400/12 - Formoterol
- Sequence 9: Formoterol - Aclidinium/Formoterol 400/6 - Aclidinium - Placebo
- Sequence 10: Placebo - Aclidinium/Formoterol 400/12 - Formoterol - Aclidinium/Formoterol 400/6
- Sequence 11: Aclidinium/Formoterol 400/6 - Formoterol - Aclidinium/Formoterol 400/12 - Placebo
- Sequence 12: Aclidinium/Formoterol 400/12 - Placebo - Aclidinium - Aclidinium/Formoterol 400/6
- Sequence 13: Aclidinium - Aclidinium/Formoterol 400/6 - Formoterol - Aclidinium/Formoterol 400/12
- Sequence 14: Formoterol - Aclidinium/Formoterol 400/12 - Placebo - Aclidinium
- Sequence 15: Placebo - Aclidinium - Aclidinium/Formoterol 400/6 - Formoterol
- Sequence 16: Aclidinium/Formoterol 400/6 - Placebo - Formoterol - Aclidinium
- Sequence 17: Aclidinium/Formoterol 400/12 - Aclidinium/Formoterol 400/6 - Placebo - Formoterol
- Sequence 18: Aclidinium - Aclidinium/Formoterol 400/12 - Aclidinium/Formoterol 400/6 - Placebo
- Sequence 19: Formoterol - Aclidinium - Aclidinium/Formoterol 400/12 - Aclidinium/Formoterol 400/6
- Sequence 20: Placebo - Formoterol - Aclidinium - Aclidinium/Formoterol 400/12
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 6 | 6 | 7 | 7 | 7 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 6 | 6 | 6 | 7
Completed | 6 | 5 | 7 | 6 | 7 | 6 | 6 | 4 | 5 | 6 | 5 | 6 | 4 | 6 | 7 | 7 | 5 | 6 | 5 | 7
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Did not meet inc/exc criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 6 | 5 | 7 | 6 | 7 | 6 | 6 | 4 | 5 | 6 | 5 | 6 | 4 | 6 | 7 | 7 | 5 | 6 | 5 | 7
Completed | 6 | 4 | 7 | 4 | 7 | 5 | 6 | 4 | 4 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 5 | 6 | 5 | 5
Not Completed | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 6 | 4 | 7 | 4 | 7 | 5 | 6 | 4 | 4 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 5 | 6 | 5 | 5
Completed | 6 | 4 | 7 | 4 | 7 | 5 | 6 | 4 | 4 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 5 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 6 | 4 | 7 | 4 | 7 | 5 | 6 | 4 | 4 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 5 | 6 | 5 | 5
Completed | 6 | 4 | 7 | 3 | 7 | 5 | 6 | 4 | 4 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: Safety population defined as all randomized patients who took at least one dose of double-blind investigational product
Arm/Group | Overall Population
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 73
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve Over 12 Hours (AUC0-12)
Time Frame: 0 to 12 hours post-dose on Day 14
Population: ITT Population defined as randomized patients who took at least one dose of double-blind investigational product and who had at least 1 baseline and 1 post-baseline assessment of FEV1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium 400 μg / Formoterol 12 μg | Aclidinium 400 μg / Formoterol 6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 78 | 83 | 82 | 75 | 81
Liters | 0.187 (0.019) | 0.189 (0.018) | 0.144 (0.018) | 0.114 (0.019) | -0.013 (0.018)
Statistical Analysis 1: Comparison: Aclidinium 400 μg / Formoterol 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Treatment and period were fixed effects, subjects was random effect, and baseline values at each period were a covariate; Least square mean difference = 0.200, 95% CI 2-sided [0.156 to 0.245], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Aclidinium 400 μg / Formoterol 6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period were fixed effects, subjects was random effect, and baseline values at each period were a covariate; Least square mean difference = 0.202, 95% CI 2-sided [0.158 to 0.245], Standard Error of Mean 0.022

2. Secondary Outcome: Change From Baseline in Morning Pre-dose (Trough) Forced Expiratory Volume in One Second (FEV1)
Time Frame: Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium 400 μg / Formoterol 12 μg | Aclidinium 400 μg / Formoterol 6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 84 | 90 | 90 | 85 | 88
Liters | 0.124 (0.018) | 0.129 (0.018) | 0.080 (0.018) | 0.071 (0.018) | -0.008 (0.018)
Statistical Analysis 1: Comparison: Aclidinium 400 μg / Formoterol 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Least square mean difference = 0.132, 95% CI 2-sided [0.083 to 0.181], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Aclidinium 400 μg / Formoterol 6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Least squares mean difference = 0.137, 95% CI 2-sided [0.088 to 0.185], Standard Error of Mean 0.025

3. Secondary Outcome: Change From Baseline in Morning Peak Forced Expiratory Volume in One Second (FEV1)
Time Frame: Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium 400 μg / Formoterol 12 μg | Aclidinium 400 μg / Formoterol 6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 84 | 90 | 90 | 85 | 87
Liters | 0.355 (0.022) | 0.348 (0.021) | 0.260 (0.021) | 0.245 (0.022) | 0.073 (0.022)
Statistical Analysis 1: Comparison: Aclidinium 400 μg / Formoterol 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Least squares mean difference = 0.281, 95% CI 2-sided [0.230 to 0.333], Standard Error of Mean 0.026
Statistical Analysis 2: Comparison: Aclidinium 400 μg / Formoterol 6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Least squares mean difference = 0.275, 95% CI 2-sided [0.224 to 0.325], Standard Error of Mean 0.026

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of investigational product, for up to 24 weeks
Arm/Group | Aclidinium 400 μg / Formoterol 12 μg | Aclidinium 400 μg / Formoterol 6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/87 | 0/91 | 1/94 | 1/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/87 | 0/91 | 0/94 | 0/92 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium 400 μg / Formoterol 12 μg (N=87) | Aclidinium 400 μg / Formoterol 6 μg (N=91) | Aclidinium 400 μg (N=94) | Formoterol 12 μg (N=92) | Placebo (N=92)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the investigator and sponsor.